CLINICAL TRIAL: NCT01901367
Title: ALL-Active: A Family-Based Lifestyle Program for Pediatric Acute Leukemia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Adam Esbenshade, Assistant Professor, Pediatric Hematology, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VICC PED 1309; P30 CA 68485 OD (Other Grant/Funding Number: National Cancer Institute); 2K12CA090625-11- A) (Other: RAC); 2K12CA090625-11 (NIH); P30CA068485 (NIH)
Record Dates: First submitted 2013-07-02; First posted 2013-07-17 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Childhood Acute Lymphoblastic Leukemia in Remission
Keywords: Adiponectin, Glucose, Insulin, Leptin
MeSH Terms: conditions — Insulin Resistance | interventions — Aftercare; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (intervention) (Experimental): Patients receive standard of care individualized diet and exercise plan and monthly booster follow-up sessions from the nutritionist and exercise physiologist and weekly phone counseling with a trained health coach to address barriers to improve plan adherence.
  Interventions: Dietary Supplement: nutritional intervention; Behavioral: exercise intervention; Other: follow-up care; Behavioral: counseling intervention; Other: quality-of-life assessment; Other: laboratory biomarker analysis; Other: questionnaire administration
- Arm II (control) (No Intervention): Patients receive standard of care individualized diet and exercise plan

INTERVENTIONS:
Dietary Supplement: nutritional intervention — Receive nutritional intervention
  Arms: Arm I (intervention)
Behavioral: exercise intervention — Receive exercise intervention
  Arms: Arm I (intervention)
Other: follow-up care — Receive booster follow-up sessions from the nutritionist and exercise physiologist
  Arms: Arm I (intervention)
Behavioral: counseling intervention — Receive phone counseling with a trained health coach
  Other Names: counseling and communications studies
  Arms: Arm I (intervention)
Other: quality-of-life assessment — Ancillary studies
  Arms: Arm I (intervention)
Other: laboratory biomarker analysis — Correlative studies
  Arms: Arm I (intervention)
Other: questionnaire administration — Ancillary studies
  Arms: Arm I (intervention)

SUMMARY:
This randomized pilot phase II trial studies how well nutritional intervention and exercise intervention works in preventing metabolic syndrome in younger patients with acute lymphoblastic leukemia. Nutritional intervention may help weight loss and improve quality of life in patients with acute lymphoblastic leukemia. Exercise may help decrease feelings of being tired caused by cancer, may help improve strength, and may help build up lost muscle tissue. Nutritional intervention plus exercise intervention may be effective at preventing metabolic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate feasibility, adherence, completion rates and participant satisfaction associated with a family based lifestyle intervention for overweight pediatric acute lymphoblastic leukemia (ALL) patients or those at high risk to become so (body mass index [BMI] >= 50th percentile).

II. Assess changes in BMI z-score, waist circumference, body composition, blood pressure exercise tolerance and physical activity at baseline, immediately post intervention and three months later.

III. Assess changes in serum glucose, insulin, leptin and adiponectin in patients over the intervention course and at 3 months post intervention.

IV. Assess changes in self-reported quality of life, physical activity, caloric intake, and fatigue associated with the nutrition and exercise program in the participant and their primary caregiver.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard of care individualized diet and exercise plan and monthly booster follow-up sessions from the nutritionist and exercise physiologist and weekly phone counseling with a trained health coach to address barriers to improve plan adherence.

ARM II: Patients receive standard of care individualized diet and exercise plan.

After completion of study treatment, patients are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pre-B cell or T cell ALL and in continuous first remission; at least 3 months into maintenance therapy with at least 7 months remaining before therapy completion
* English speaking patient and primary caregiver
* BMI >= 75th percentile at time of study enrollment; (patients >= 75th percentile were selected as they were the group in our preliminary data that had a high risk of becoming overweight during maintenance therapy)
* Provision of informed consent by primary caregiver

Exclusion Criteria:

* Any physical or mental limitation that would prevent participation in study activities (Including but not limited to grade 4 neuropathy or inability to ambulate)
* As this is intended to be a family-based intervention, all family members will be invited to participate, including those living in more than one household, however endpoints will only be assessed formally in the patient and identified primary caregiver; siblings are not required for participation.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2013-05; Primary Completion 2014-09-30 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Percentage change in number of pediatric ALL patients with BMI ≥ 75th percentile who agree to be randomized to participate in a lifestyle intervention program. | Baseline and at 6 months
  Patients undergo a nutrition and counseling intervention designed to decrease their calorie intake, meet micronutrient recommendations, and participate in an exercise plan. Feasibility is defined as >50% of patients who complete the intervention

SECONDARY OUTCOMES:
Percentage of increase or decrease in BMI of pediatric ALL patients with a BMI > 75th percentile who undergo a nutrition and counseling intervention compared to a control group of pediatric ALL patients who do not undergo intervention | At 3 months and at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Adam Esbenshade, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States